CLINICAL TRIAL: NCT01505192
Title: Determination of the Physiological Reference Values of Trend of Hemoglobin in the Post-partum Period After Spontaneous Vaginal Delivery. A Sequential Pilot Study Using the Noninvasive Continuous Technology of SpHb
Brief Title: Noninvasive Continuous Measurement of SpHb After Spontaneous Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Città di Roma Hospital (Other)
Responsible Party: Principal Investigator, Silvia Stirparo, Staff Anesthesiologist, Città di Roma Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Postpartum non invasive Hb
Record Dates: First submitted 2011-12-28; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Delivery Uterine
Keywords: Those in Labor, Delivery and the Puerperium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: continuous Hb monitor — Pre and post partum non invasive continuous Hb monitor
  Other Names: Masimo Radical 7

SUMMARY:
Aim of this study is to determine the physiological reference individual values (RI) of maternal continuous SpHb immediately after delivery in the post-partum period (continuous monitoring up to 2 hours after delivery) in order to establish the physiological Hb variations in response to the physiological blood loss due to delivery.

During labor all parturients will be tested for standard Laboratory Hb and monitored for at least 30 minutes with SpHb monitoring equipment (Radical-7™ Pulse CO-Oximeter and Rainbow DiSposable™ Adult Adhesive Sensor), and these values will be considered to be the baseline values.

Immediately after spontaneous vaginal delivery, venous blood sample will be taken for Hb determination and Radical 7 equipment for SpHb will be connected to the patient's finger and will be recorded for at least two hours after delivery. At the end of this period of observation a venous blood sample will be taken for Hb determination. Additional measurements of both SpHb and Lab Hb will be performed 24 hours after delivery.

DETAILED DESCRIPTION:
Background and Significance:

Pregnancy and childbirth involve health risks, even for women without any pre-existing health problems. Postpartum hemorrhage is one of most common complications for delivering mothers and causes 19% of in-hospital maternal deaths (Bateman BT et al. "The Epidemiology of Postpartum Hemorrhage in a Large, Nationwide Sample of Deliveries" Anesthesia and Analgesia 2010 110:1368-1373) . Due to pregnancy physiological changes, maternal bleeding is typically discovered after a significant change in vital signs, and/or symptoms, and usually confirmed with an invasive laboratory hemoglobin test. This can result in late detection of bleeding that can affect patient outcome. Early detection of signs and symptoms of obstetric hemorrhage is therefore crucial. Non-invasive and continuous hemoglobin (SpHb) monitoring system quickly measures current hemoglobin levels and continuously tracks them in real-time to detect falling hemoglobin levels that may, in turn, represent an early sign of a potential hemorrhage. Unfortunately there is no validation of the clinical accuracy of the Rainbow device for the noninvasive and continuous hemoglobin (SpHb) monitoring in the obstetric setting nor any information concerning its use as a tool for the early detection of postpartum hemorrhage.

The investigators therefore propose to undertake an open, preliminary, sequential pilot study to determine the physiological values (RI) of maternal continuous SpHb in the post-partum period.

Study Objective:

To determine the physiological reference individual values (RI) of maternal continuous SpHb immediately after delivery in the post-partum period (continuous monitoring up to 2 hours after delivery) in order to establish the physiological Hb variations in response to the physiological blood loss due to delivery.

Inclusion and exclusion criteria

Healthy parturients in labor will be asked to be enrolled in the study and informed consent will be obtained.Parturients will be consecutively included in this study. Bleeding risk subjects will be excluded (parturients who had:

Operative or instrumental vaginal delivery,Estimated blood loss greater than 500 mL, who had II and III degree perineal lacerations, any coagulation disorder or anticoagulant therapy)

Sample Size Since we have no available information on the expected distribution of the outcome, we will use a sequential design. The main endpoint of our analysis will be a reliable estimate for the outcome expected in healthy women after labor.

The investigators will state their target estimate as being reliable when the ratio between the estimate and its standard error is smaller than 2.

The International Federation of Clinical Chemistry (IFCC) and Clinical Laboratory and Standards Institute (CLSI) guidelines in 2008 recommended to establish RIs with at least 120 reference individuals using the nonparametric ranking method (Clinical and Laboratory Standards Institute. Defining, Establishing, and Verifying Reference Intervals in the Clinical Laboratory; Approved Guideline. 3rd ed. Wayne, PA: CLSI; 2008) and thus we will include in the study a sample of at least 120.

Methods During labor all parturients will be tested for standard Laboratory Hb and monitored for at least 30 minutes with SpHb monitoring equipment (Radical-7™ Pulse CO-Oximeter and Rainbow DiSposable™ Adult Adhesive Sensor), and these values will be considered to be the baseline values.

Immediately after spontaneous vaginal delivery, venous blood sample will be taken for Hb determination and Radical 7 equipment for SpHb will be connected to the patient's finger and will be recorded for at least two hours after delivery. At the end of this period of observation a venous blood sample will be taken for Hb determination. Additional measurements of both SpHb and Lab Hb will be performed 24 hours after delivery.

According to the SpHB data collection-research protocol, sensor site will be connected to the patient's ring finger of the non-dominant hand. Sensor handling and placement will also follow the instructions of the SpHB data collection-research protocol.

Sensor will be attached to the same arm as the blood draw. Sensor placement on the hand of the side with the blood pressure cuff will be avoided unless they are drawing blood from that extremity. Placing the sensor and drawing blood from the same arm that is being used for IV infusions will be also avoided.

SpHb results will be not included when the Perfusion Index (PI, noninvasive index of peripheral perfusion and vasomotor tone) values will be less than 0.5.

Concerning blood sampling, blood will be drawn directly into the vacutainer by using a needle no smaller than 20G and analyzed within 15 min of the blood draw.

In Vivo adjustment and Trend Accuracy

SpHb accuracy with an in vivo adjustment will be calculated by using the new Radical 7 equipment with in vivo adjustment feature software which will take the bias between the first SpHb and first laboratory tHb measurement and will adjust all subsequent measurements for that case.

The trend accuracy will be calculated by using the following time points: pre-delivery, 2 hrs after delivery and 24 hr after delivery.

Calibrated SpHb measurements will be compared to subsequent laboratory values to create a Bland Altman plot and calculate bias, and confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy parturients in labor

Exclusion Criteria:

* Parturient with coagulation defects, or with anticoagulant therapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-03 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
SpHb monitoring equipment (Radical-7™ Pulse CO-Oximeter and Rainbow DiSposable™ Adult Adhesive Sensor, Masimo, Irvine, CA. Continuous Hemoglobin evaluation, measure unit: g/dL | 24 hours postpartum
  To determine the physiological reference individual values (RI) of maternal continuous SpHb immediately after delivery in the post-partum period (continuous monitoring up to 2 hours after delivery) in order to establish the physiological Hb variations in response to the physiological blood loss due to delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stirparo, MD, Principal Investigator — Città di Roma Hospital; Giorgio Capogna, MD, Study Chair — Cittàdi Roma Hospital
Locations (1):
- Città di Roma Hospital, Roma, Italy